CLINICAL TRIAL: NCT03039972
Title: Prospective Evaluation of Changes in Renal Function and Body Composition in Patients With Pulmonary Hypertension
Brief Title: Changes in Renal Function and Body Composition in Pulmonary Hypertension
Status: Completed | Type: Observational
Sponsor: University of Giessen (Other)
Responsible Party: Principal Investigator, Faeq Husain, Senior Physician Nephrology, University of Giessen
Other Study IDs: AZ 239/16
Record Dates: First submitted 2017-01-29; First posted 2017-02-01 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Pulmonary Hypertension; Renal Function Abnormal
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Collection of only residual material (blood, urine) for Deutsche Zentrum für Lungenforschung Biobank.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pulmonary Hypertension: Adult outpatients with suspected or prediagnosed pulmonary hypertension irrespective of subclass and all chronic kidney disease stages
  Interventions: Diagnostic Test: No intervention

INTERVENTIONS:
Diagnostic Test: No intervention — No intervention

SUMMARY:
Changes in renal function and body composition in patients with pulmonary hypertension

DETAILED DESCRIPTION:
This prospective single-center study is designed to analyze changes in renal function and body composition in patients with suspected or pre-diagnosed pulmonary hypertension at pulmonary hypertension outpatient clinic, University Hospital Giessen and Marburg, Campus Giessen.

ELIGIBILITY:
Inclusion Criteria:

* Subjects older than 18 years at pulmonary hypertension outpatient clinic
* Subjects who signed informed consent forms

Exclusion Criteria:

* Patients refusing to participate or withdraw consent during follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with suspected or pre-diagnosed pulmonary hypertension at pulmonary hypertension outpatient clinic, University Hospital Giessen and Marburg, Campus Giessen
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2017-01-25 (Actual); Primary Completion 2019-10-07 (Actual); Study Completion 2020-07-09 (Actual)

PRIMARY OUTCOMES:
Changes in renal function in patients with pulmonary hypertension | 1 year
  Estimated GFR based on Chronic Kidney Disease Epidemiology Collaboration-creatinine-cystatin C will be used to determine renal function at baseline and at 1 year follow-up

SECONDARY OUTCOMES:
Changes in hydration status in patients with pulmonary hypertension | 1 year
  Bioimpedance analysis will be used to determine hydration status at baseline and at 1 year follow-up
Changes in nutritional status in patients with pulmonary hypertension | 1 year
  Bioimpedance analysis will be used to determine lean tissue and fat mass at baseline and at 1 year follow-up
Prognostic value of baseline renal function, hydration and nutritional status on pulmonary hypertension-associated morbidity and mortality | 1 year
  pulmonary hypertension-associated morbidity and mortality (defined as escalation of pulmonary hypertension-specific therapy, unscheduled hospitalization and all-cause mortality) will be prospectively assessed during follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Werner Seeger, MD, Study Director — Department of Internal Medicine II, Division of Pulmonology, Nephrology and Critical Care Medicine
Locations (1):
- University Clinic Giessen and Marburg - Campus Giessen, Giessen, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, ICF
Time Frame: Starting 6 months after publication

REFERENCES:
- [Background] Bellomo R, Prowle JR, Echeverri JE. Diuretic therapy in fluid-overloaded and heart failure patients. Contrib Nephrol. 2010;164:153-163. doi: 10.1159/000313728. Epub 2010 Apr 20. PMID 20428001
- [Background] Ronco C, Verger C, Crepaldi C, Pham J, De Los Rios T, Gauly A, Wabel P, Van Biesen W; IPOD-PD Study Group. Baseline hydration status in incident peritoneal dialysis patients: the initiative of patient outcomes in dialysis (IPOD-PD study)dagger. Nephrol Dial Transplant. 2015 May;30(5):849-58. doi: 10.1093/ndt/gfv013. Epub 2015 Mar 11. PMID 25762355
- [Result] Navaneethan SD, Wehbe E, Heresi GA, Gaur V, Minai OA, Arrigain S, Nally JV Jr, Schold JD, Rahman M, Dweik RA. Presence and outcomes of kidney disease in patients with pulmonary hypertension. Clin J Am Soc Nephrol. 2014 May;9(5):855-63. doi: 10.2215/CJN.10191013. Epub 2014 Feb 27. PMID 24578332
- [Result] Damman K, van Deursen VM, Navis G, Voors AA, van Veldhuisen DJ, Hillege HL. Increased central venous pressure is associated with impaired renal function and mortality in a broad spectrum of patients with cardiovascular disease. J Am Coll Cardiol. 2009 Feb 17;53(7):582-588. doi: 10.1016/j.jacc.2008.08.080. PMID 19215832